CLINICAL TRIAL: NCT01845454
Title: A Dose-Optimization Study for the Initial Treatment of Dysplastic Barrett's Esophagus With trūFreeze™ Spray Cryotherapy ("DOSE" Trial)
Brief Title: A Dose-Optimization Study for the Initial Treatment of Dysplastic Barrett's Esophagus With trūFreeze™ Spray Cryotherapy
Acronym: DOSE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: poor enrollment and study design
Sponsor: CSA Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 006
Record Dates: First submitted 2013-04-25; First posted 2013-05-03 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: Barrett's Esophagus
Keywords: Barrett's Esophagus; Spray cryotherapy
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dose 1 (Active Comparator): The first 15 patients enrolled will receive a dose of 1 application of 20 seconds each of spray cryotherapy using the trūFreeze™ spray cryotherapy device throughout the affected tissue.
  Interventions: Device: trūFreeze™ Spray Cryotherapy
- Dose 2 (Active Comparator): If a second cohort of 15 participants is necessary, the next dose will include 1 application of 30 seconds each of spray cryotherapy using the trūFreeze™ spray cryotherapy device throughout the affected tissue.
  Interventions: Device: trūFreeze™ Spray Cryotherapy
- Dose 3 (Active Comparator): If an additional cohort of 15 participants is necessary, the next dose will include 2 applications of 20 seconds each of spray cryotherapy using the trūFreeze™ spray cryotherapy device throughout the affected tissue.
  Interventions: Device: trūFreeze™ Spray Cryotherapy
- Dose 4 (Active Comparator): If an additional cohort of 15 participants is necessary, the next dose will include 2 applications of 30 seconds each of spray cryotherapy using the trūFreeze™ spray cryotherapy device throughout the affected tissue.
  Interventions: Device: trūFreeze™ Spray Cryotherapy

INTERVENTIONS:
Device: trūFreeze™ Spray Cryotherapy — The trūFreeze™ System consists of a console containing a holding tank for medical grade liquid nitrogen and a spray tip CSATM Catheter. The physician uses the console to initiate and control the flow and duration of the cryogen spray. The liquid nitrogen is propelled through a spray CSATM Catheter to the selected site by pressure in the holding tank and freezing techniques are monitored by direct visualization with an endoscope. Once the freezing is completed, the cryogen flow is terminated and the thawing system may be engaged to allow accessory removal. If multiple cycles are used, thawing is initiated at the end of the procedure.

SUMMARY:
The primary objective of this study is to determine the percentage segment regression after spray cryotherapy in a dose-escalation study performed in patients with dysplastic Barrett's Esophagus (BE) using trūFreeze™ spray cryotherapy within the currently recommended therapeutic range.

Secondary objectives are the determination of safety related outcomes such as esophageal stricture.

DETAILED DESCRIPTION:
This is an adaptive dose-escalation clinical trial using trūFreeze™ spray cryotherapy for the treatment of dysplastic Barrett's Esophagus in a clinical setting.

Participants will be enrolled in cohorts of up to 15. Each cohort will receive a similarly dosed spray cryotherapy treatment, based on outcomes from the previous cohort. Participants will receive one treatment with spray cryotherapy per the protocol and will then be followed clinically. During the next scheduled clinical endoscopy, participants will be assessed for percent regression of disease following the spray cryotherapy treatment. A determination will be made regarding effectiveness of each dose based on the number of subjects that achieve the primary outcome criterion (>= 50 percent BE segment regression).

The first cohort of up to 15 participants will receive an upper endoscopy in which systematic images of the esophagus will be taken for the research study and will then receive a treatment with spray cryotherapy using the trūFreeze™ system. These participants will have a clinical follow-up endoscopy scheduled approximately 2 months after the initial spray cryotherapy procedure. During the follow-up endoscopy, physicians will be asked to provide an estimate of the percent regression of disease as well as systematic images of the esophagus. These images will be sent to a central panel of masked experts who will assess percent regression of disease compared to images taken prior to the first ablation procedure.

Interim reviews of potential dose effectiveness will occur when 7 and 11 participants have completed the follow-up visit. If during an interim review at least 5 participants experience a sub-therapeutic response, the dose will be considered sub-therapeutic as not meeting the definition of "fully effective," the cohort will be closed to new enrollment, and enrollment on a new cohort at the next higher dose will begin. If during an interim review less than 5 participants experience a sub-therapeutic response, enrollment on that cohort will continue.

If/when enrollment on a cohort reaches 15 participants a decision will be made regarding the effectiveness of the dose. If a dose is found to be "ineffective" or "partially effective," then a new cohort of individuals will be enrolled at a prescribed higher starting dose. If a dose is found to be "fully effective," then a confirmatory cohort will be enrolled at the same dose to confirm results. Enrollment will continue until a "fully effective" therapeutic dose of spray cryotherapy is identified and confirmed in two cohorts of 15 participants each.

ELIGIBILITY:
Inclusion Criteria:

* English speaking males or females aged 18 to 80 who are candidates for sedated endoscopy with treatment of BE.
* At least 3 centimeters segment length of Barrett's Esophagus (BE) with or without circumferential involvement (i.e. CxM3) and with high grade or low grade dysplasia based on pathology results from 4 quadrant biopsies taken every 1-2 centimeter throughout the BE. All readings of dysplasia will be confirmed by an expert pathologist.
* Willing to undergo spray cryotherapy and judged by patient's physician as an appropriate candidate for this therapy.
* Able to read, comprehend, and complete the informed consent form

Exclusion Criteria:

* Bleeding disorder or other contraindication of spray cryotherapy.
* History of partial or complete esophagectomy.
* Current or past diagnosis of invasive esophageal cancer (previous intramucosal cancer is allowable, if removed by endoscopic mucosal resection with histologically confirmed negative lateral and deep margins).
* Pregnant women
* Contraindication to endoscopic spray cryotherapy as outlined in the directions for use for the device
* Previous endoscopic ablation treatment (such as radiofrequency ablation (RFA) or photodynamic therapy (PDT)).
* Previous chest external beam radiation therapy.
* Previous wide-area endoscopic resection or submucosal dissection. Previous focal mucosal resection is permitted (maximum 2 previous EMR's of 2cm or less removed representing less than 25% of the circumference of the esophagus removed).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-04; Primary Completion 2014-11 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of Spray Cryotherapy Dose: Percent Regression of Disease Following Baseline Spray Cryotherapy | Next follow-up endoscopy scheduled as routine care (2 months +/- 4 weeks)
  Percent regression of disease will be used to determine efficacy of spray cryotherapy dose used. If at follow-up there is less than a 50% reduction in Barrett's Esophagus, the outcome will be characterized as sub-therapeutic for that participant. If a 50% or greater reduction is seen then this would be characterized as therapeutic. In each cohort of 15:
  * If less than 5 subjects are found to have a "therapeutic" response , dose = "ineffective"
  * If 5 to 10 subjects are found to have a "therapeutic" response, dose = "partially effective"
  * If 11 to 15 subjects have a "therapeutic" response, dose = "fully effective"
  If a dose is found to be "ineffective" or "partially effective", then a new evaluation cohort of 15 individuals will be enrolled on the next higher dose. If the dose is considered "fully effective" then a second cohort of 15 individuals will be enrolled on the same dose to confirm. Enrollment continues until a fully effective dose is attained and confirmed

SECONDARY OUTCOMES:
Safety Outcomes | Next follow-up endoscopy scheduled as routine care (2 months +/- 4 weeks)
  Secondary objectives are the determination of safety related outcomes such as esophageal stricture and will be captured by reportable events.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Shaheen, MD, MPH, Principal Investigator — UNC Chapel Hill
Locations (6):
- United States (6):
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - University of Maryland, Baltimore, Maryland
  - Columbia University, New York, New York
  - University of North Carolina, Chapel Hill, Chapel Hil, North Carolina
  - Ahuja/University Hospitals, Beachwood, Ohio
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No